CLINICAL TRIAL: NCT00699231
Title: Study to Evaluate the Immunogenicity, Reactogenicity and Safety of GSK Biologicals' (Previously SmithKline Beecham Biologicals') MPL-Adjuvanted Recombinant Hepatitis B Vaccine Versus Engerix™-B, in Haemodialysis Patients
Brief Title: Evaluation of Immunogenicity, Reactogenicity and Safety of HBV-MPL Vaccine vs Engerix™-B, in Haemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208129/002
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant hepatitis B vaccine; Adjuvant
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Group A1 (Active Comparator): Non-responders to vaccination after at least 7 previous injections
  Interventions: Biological: Engerix™-B
- Group A2 (Experimental): Non-responders to vaccination after at least 7 previous injections
  Interventions: Biological: HBV-MPL vaccine 208129
- Group B1 (Active Comparator): Vaccine-responders requiring a booster dose
  Interventions: Biological: Engerix™-B
- Group B2 (Experimental): Vaccine-responders requiring a booster dose
  Interventions: Biological: HBV-MPL vaccine 208129
- Group C1 (Active Comparator): Volunteers participating in the hospital's vaccination program
  Interventions: Biological: Engerix™-B
- Group C2 (Experimental): Volunteers participating in the hospital's vaccination program
  Interventions: Biological: HBV-MPL vaccine 208129
- Group D1 (Active Comparator): Unvaccinated haemodialysis patients
  Interventions: Biological: Engerix™-B
- Group D2 (Experimental): Unvaccinated haemodialysis patients
  Interventions: Biological: HBV-MPL vaccine 208129

INTERVENTIONS:
Biological: HBV-MPL vaccine 208129 — IM injection
  Arms: Group A2; Group B2; Group C2; Group D2
Biological: Engerix™-B — IM injection
  Arms: Group A1; Group B1; Group C1; Group D1

SUMMARY:
This trial is designed to evaluate the immunogenicity, reactogenicity and safety of an MPL-adjuvanted recombinant hepatitis B vaccine in comparison with those of Engerix™-B in haemodialysis patients with or without previous vaccination against hepatitis B

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Dialysis patients
* A medical examination including physical examination and medical history as well as serological screening established acceptability for enrollment into the study.
* Age: from 18 years onwards
* Seronegative for anti- hepatitis antibodies

Exclusion Criteria:

* History of persistent hepatic, cardiac or respiratory disease
* Any acute disease at the moment of entry into the study
* Chronic alcohol consumption
* Hepatomegaly, right upper quadrant pain or tenderness
* Any treatment with coticosteroids or immunomodulating drugs
* Known hypersensitivity to any component of the vaccine
* Simultaneous participation in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1992-02; Primary Completion 1992-12 (Actual); Study Completion 1992-12 (Actual)

PRIMARY OUTCOMES:
Occurrence and intensity of solicited local and general symptoms | 4-day follow-up period after each vaccination
Occurrence of unsolicited adverse events | During the course of the study
Occurrence of serious adverse events | During the course of the study
Anti-HBs antibody concentrations | Pre, Day 0, Day 30, Day 60, Day 90, Day 120, D180, D210 depending on group allocation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Brussels, Belgium